CLINICAL TRIAL: NCT03108456
Title: Evaluation of Treatment Strategies for Severe CaLcIfic Coronary Arteries: Orbital Atherectomy vs. Conventional Angioplasty Technique Prior to Implantation of Drug-Eluting StEnts: The ECLIPSE Trial
Acronym: ECLIPSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-0011-P
Record Dates: First submitted 2017-02-17; First posted 2017-04-11 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease; Non ST Segment Elevation Myocardial Infarction
Keywords: atherectomy; CAD; severe calcium; orbital atherectomy; minimum stent area
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Orbital Atherectomy (OA) (Active Comparator): The Diamondback 360® Coronary Orbital Atherectomy System (OAS) will be used for orbital atherectomy (OA) vessel preparation prior to implantation of a drug-eluting stent.
  Interventions: Device: Orbital Atherectomy
- Conventional Balloon Angioplasty (Active Comparator): Coronary balloons cleared or approved for commercial use by the Food and Drug Administration will be used for conventional balloon angioplasty prior to implantation of a drug-eluting stent.
  Interventions: Device: Balloon

INTERVENTIONS:
Device: Orbital Atherectomy — Vessel preparation with Orbital Atherectomy followed by balloon pre-dilatation
  Arms: Orbital Atherectomy (OA)
Device: Balloon — Vessel preparation with conventional and/or specialty balloons
  Arms: Conventional Balloon Angioplasty

SUMMARY:
This trial will evaluate Orbital Atherectomy compared to conventional balloon angioplasty technique for the treatment of severely calcified lesions prior to implantation of drug-eluting stents (DES).

ELIGIBILITY:
General Inclusion Criteria:

1. Subject is 18 years of age or older.
2. Subject presents with:

   1. stable ischemic heart disease or
   2. acute coronary syndrome (NSTEMI or unstable angina), or
   3. stabilized recent STEMI (>48 hours prior to randomization procedure)
3. Subject has signed the Institutional Review Board (IRB) or Ethics Committee (EC) approved ECLIPSE trial Informed Consent Form (ICF) prior to any trial related procedures.

General Exclusion Criteria

1. Subject has a history of any cognitive or mental health status that would interfere with trial participation.
2. Subject is participating in or has plans to participate in any other investigational drug or device trial that has not reached its primary endpoint.
3. Subject is a female who is pregnant.
4. Subject is receiving or scheduled to receive chemotherapy within thirty (30) days prior or any time after the randomization procedure.
5. Subject has a life expectancy of ≤ 12 months.
6. Subject has undergone any prior PCI in the target vessel or its branches 12 months prior to randomization.
7. Subject has undergone a PCI procedure that is unsuccessful or with complications within 30 days prior to randomization, including during the randomization procedure.
8. Any cardiac intervention or cardiac surgery planned within 12 months post randomization procedure aside from a potential planned staged PCI as part of the randomized treatment strategy.
9. Subject has major valve disease and underwent intervention within 30 days prior to randomization.
10. Subject has received a heart transplant.
11. Evidence of heart failure by at least one of the following (heart failure assessment is not required per protocol but must be reviewed prior to enrollment if data is available):

    1. Most recent LVEF ≤25%, or
    2. Current heart failure defined as dyspnea at rest (NYHA class IV assessed day of procedure), or
    3. Killip class ≥2 (post STEMI patients)
12. Planned use in the randomized lesion(s) of a bare metal stent (BMS), bioresorbable scaffold (BRS), non-stent treatment only.
13. Subject has a known sensitivity to contrast media, which cannot be adequately pre-medicated.
14. Subject has a relative or absolute contraindication to dual antiplatelet therapy or (for patients with atrial fibrillation) single antiplatelet therapy (P2Y12 inhibitor preferred) with an anticoagulant for at least 6 months after PCI.
15. Subject has a history of a stroke or transient ischemic attack (TIA) within six (6) months prior to randomization, or any permanent neurologic deficit.
16. Subject has a history of bleeding diathesis or coagulopathy or intention to refuse blood transfusion if one should become necessary.
17. Subject has evidence of an active infection on the day of the randomization procedure requiring oral or intravenous antibiotics.
18. Subject with known allergy to atherectomy lubricant components including soybean oil, egg yolk phospholipids, glycerin and sodium hydroxide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2005 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2024-06-12 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Acute Minimum Stent Area (MSA) | Procedure
  In-stent minimal cross-sectional area as assessed by optical coherence tomography (OCT) at the conclusion of the procedure in the OCT imaging cohort.
Target Vessel Failure (TVF) | 1-Year
  Target vessel failure, defined as the composite of cardiac death, target vessel related myocardial infarction (MI), or ischemia-driven target vessel revascularization.

SECONDARY OUTCOMES:
Procedural Success | Procedure
  Procedural success, defined as successful stent delivery with final Core Lab defined Thrombolysis in Myocardial Infarction (TIMI) flow three (3) and angiographic in-stent diameter stenosis (DS) ≤20%, and with the absence of any of the following: stent loss, coronary perforation, or intra-procedural death.
Strategy Success | Procedure
  Strategy success, defined as procedural success without crossover to alternative treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Kirtane, MD, SM, Principal Investigator — Columbia University Medical Center / New York-Presbyterian Hospital; Philippe Généreux, MD, Principal Investigator — Morristown Medical Center
Locations (104):
- United States (104):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Mercy Gilbert Medical Center, Chandler, Arizona
  - St. Luke's Medical Center, Phoenix, Arizona
  - Arizona Heart Hospital, Phoenix, Arizona
  - Yavapai Regional Medical Center, Prescott, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - University of California - San Diego, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - San Francisco VA Medical Center, San Francisco, California
  - Denver VA Medical Center, Denver, Colorado
  - Colorado Heart and Vascular, Lakewood, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - The Cardiac & Vascular Institute Research Foundation, Gainesville, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Heart Institute at Largo, Largo, Florida
  - AdventHealth Ocala, Ocala, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Palm Beach Gardens Medical Center, Palm Beach Gardens, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - University of Illinos - Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Indiana University, Indianapolis, Indiana
  - St. Vincent Heart of Indiana, Indianapolis, Indiana
  - Community Hospital, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - Iowa Heart Center, West Des Moines, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - U of L Health, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Lafayette General Medical Center, Lafayette, Louisiana
  - Ochsner Medical, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Detroit Medical Center, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital and Medical Center, Detroit, Michigan
  - Metropolitan Cardiology Consultants, Coon Rapids, Minnesota
  - Essentia Health, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - Forrest General - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Stern Cardiovascular, Southaven, Mississippi
  - VA St. Louis Healthcare System, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - St. Louis University, St Louis, Missouri
  - Deborah Heart and Lung Medical Center, Browns Mills, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - St. Peter's Hospital, Albany, New York
  - New York University School of Medicine, New York, New York
  - Columbia University Medical Center / New York-Presbyterian Hospital, New York, New York
  - Northwell Health, New York, New York
  - Hudson Valley Cardiovascular Practice, PC, Poughkeepsie, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore-Einstein Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Mercy Health West Hospital, Cincinnati, Ohio
  - University Hospital Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Riverside Methodist Hospital/Ohio Health, Columbus, Ohio
  - Premier Health Specialists, Dayton, Ohio
  - Oklahoma Heart Hospital - South Campus, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - St. John's Health System, Tulsa, Oklahoma
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Sanford Heart Hospital, Sioux Falls, South Dakota
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Methodist Health, Dallas, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Sentara Cardiovascular, Norfolk, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Genereux P, Kirtane AJ, Kandzari DE, Armstrong EJ, Krucoff MW, Redfors B, Ben-Yehuda O, Lerew DR, Ali ZA, Maehara A, O'Neill WW, Stone GW. Randomized evaluation of vessel preparation with orbital atherectomy prior to drug-eluting stent implantation in severely calcified coronary artery lesions: Design and rationale of the ECLIPSE trial. Am Heart J. 2022 Jul;249:1-11. doi: 10.1016/j.ahj.2022.03.003. Epub 2022 Mar 12. PMID 35288105
- [Derived] Maehara A, Kirtane AJ, Genereux P, Matsumura M, Lewis BE, Shlofmitz RA, Dohad S, Choudary J, Dahle T, Pineda AM, Shunk KA, Popma A, Redfors B, Ali ZA, Krucoff MW, Armstrong EJ, Kandzari DE, Phalakornkule K, Kraemer C, Stiefel KM, Jones DE, Buccola JR, Chambers JW, Stone GW. Calcium Modification After Orbital Atherectomy and Balloon Angioplasty in Severely Calcified Lesions: The ECLIPSE OCT Substudy. Circ Cardiovasc Interv. 2026 Jan;19(1):e015588. doi: 10.1161/CIRCINTERVENTIONS.125.015588. Epub 2025 Dec 3. PMID 41332372
- [Derived] Kirtane AJ, Genereux P, Lewis B, Shlofmitz RA, Dohad S, Choudary J, Dahle T, Pineda AM, Shunk K, Maehara A, Popma A, Redfors B, Ali ZA, Krucoff M, Armstrong E, Kandzari DE, O'Neill W, Kraemer C, Stiefel KM, Jones DE, Chambers J, Stone GW; ECLIPSE Investigators. Orbital atherectomy versus balloon angioplasty before drug-eluting stent implantation in severely calcified lesions eligible for both treatment strategies (ECLIPSE): a multicentre, open-label, randomised trial. Lancet. 2025 Apr 12;405(10486):1240-1251. doi: 10.1016/S0140-6736(25)00450-7. Epub 2025 Mar 30. PMID 40174596